CLINICAL TRIAL: NCT05999357
Title: A Phase II Study evaluaTing intRacranial effIcacy of JDQ443 in patiEnts With KRAS G12C+ NSCLC and bRain Metastases
Brief Title: JDQ443 for KRAS G12C NSCLC Brain Metastases
Acronym: STRIDER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis discontinued develpment of JDQ443
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CJDQ443B1NL01T; 2023-505721-13-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-08-02; First posted 2023-08-21 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Brain Metastases, Adult; KRAS G12C
Keywords: non small cell lung cancer; brain metastases; KRAS G12C; JDQ443
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — JDQ443

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, 2-cohort phase II study. Cohort A: asymptomatic, untreated BM, Cohort B: asymptomatic, treated BM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adult patients with KRAS G12C+ NSCLC and brain metastases (Experimental): Cohort A: adult patients with KRAS G12C+ NSCLC and untreated asymptomatic BM Cohort B: Adult patients with KRAS G12C+ NSCLC and treated asymptomatic BM
  JDQ443 200 mg BID until unacceptable toxicity or disease progression
  Interventions: Drug: JDQ443

INTERVENTIONS:
Drug: JDQ443 — JDQ443 tablets, orally administered
  Other Names: no other name

SUMMARY:
The goal of this phase II clinical trial is to evaluate the intracranial efficacy of JDQ443, a KRAS G12C inhibitor in patients with KRAS G12C+ NSCLC and brain metastases (cohort A: asymptomatic, untreated brain metastases, cohort B: asymptomatic, treated brain metastases). The main question it aims to answer is to evaluate the intracranial efficacy, according to RANO-BM criteria, in patients with asymptomatic and untreated brain metastases.

Participants will receive JDQ443 200 mg BID until unacceptable toxicity or disease progression.

DETAILED DESCRIPTION:
In the past decade, the treatment and prognosis of patients with metastatic non-small cell lung cancer (NSCLC) has significantly improved, due to new systemic treatments (i.e. intravenous or oral therapy). NSCLC is increasingly subtyped based on the presence of certain mutations in the NSCLC for which targeted therapies have become available. KRAS G12C is the most commonly found mutation, and recently oral therapies (sotorasib in the EU and USA, adagrasib in the USA) have become available.

Brain metastasis (BM) incidence in patients with KRAS G12C+ non-small cell lung cancer (NSCLC) is high, but unfortunately, except for one small trial with adagrasib, patients with BM were excluded from most clinical trials with KRAS G12C inhibitors. Furthermore, sotorasib is not very well able to reach the central nervous system (CNS). Adagrasib can penetrate into the CNS, but this comes with relevant treatment related toxicity (mainly gastro-intestinal and liver). JDQ443 is a new oral KRAS G12C inhibitor, that preclinically has the same ability as adagrasib to reach the CNS, but based on small series seems to have less toxicity. As toxicity seems favourable for JDQ443 compared with sotorasib and adagrasib, and as preclinically, CNS penetration seems comparable to adagrasib, data regarding the efficacy of JDQ443 on BM is urgently needed. Therefore the main objective of this trial is to evaluate the intracranial efficacy of JDQ443 in patients with KRAS G12C+ NSCLC and asymptomatic untreated BM. Furthermore, there will be an exploratory cohort for patients with asymptomatic and treated BM.

The intervention consists of JDQ443 200 mg BID until unacceptable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Participant is an adult ≥ 18 years of age at the time of informed consent.
3. ECOG performance status ≤2.
4. Estimated life expectancy of 12 weeks or more
5. Metastatic (stage IV) NSCLC with the presence of a KRAS G12C mutation (local test, tissue as well as liquid biopsy allowed) and untreated or progressing asymptomatic BM (cohort A) or treated and stable BM (cohort B).
6. BM not in eloquent area (all patients have at least to be discussed with a neurologist, and preferably they are discussed in a neuro-oncology MDT). If treated with radiotherapy and stable, these patients are eligible for cohort B.
7. Max BM size 2 cm in longest diameter (for each BM) for cohort A
8. For cohort A: at least one untreated brain metastasis ≥ 5mm:

   1. Patients with largest measurable intracranial lesion ≥5 mm but <10 mm may be allowed to enroll upon agreement with the principal investigator (for patients with target lesions of ≥ 5mm but <10 mm, 1.5 mm slice thickness brain MRI is required).
   2. Prior local treatment is permissible if completed at least 14 days prior to study enrollment and provided unequivocal progression in the lesion has since occurred or if new lesions have occurred.
   3. For at least 7 days prior to first dose of JDQ443 in this study: Patient must be asymptomatic from CNS metastases and on a stable dose of corticosteroids, with a maximum of 4 mg dexamethasone/day. Anti-epileptic dose should also be stable for 7 days.
9. Participant must have recovered from all toxicities related to prior treatments to grade ≤ 1 (CTCAE v 5.0). Exception to this criterion are alopecia and vitiligo of any grades.
10. Adequate organ function including the following laboratory values at the screening visit:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (without growth factor support),
    * Platelets ≥ 100 x 109/L (without growth factor support),
    * Hemoglobin (Hgb) ≥ 6 mmol/l (= 9 g/dl) (7 days without transfusions or growth factor support),
    * Aspartate transaminase (AST) ≤ 3 x ULN,
    * Alanine transaminase (ALT) ≤ 3 x ULN,
    * Total bilirubin ≤ 1.5 ULN,
    * Serum lipase ≤ 1.5 x ULN,
    * Creatinine clearance ≥ 60 mL/min by calculation using Cockcroft-Gault formula or based on 24-hour urine sample assessment.
11. Participant is capable of swallowing study medication and following instructions regarding study treatment administration.
12. Participant must be able to communicate with the Investigator and comply with the requirements of the study procedures.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Leptomeningeal metastasis (based on MRI or CSF cytology, if strong suspicion despite negative MRI, CSF analysis should be done)
2. Previous treatment with KRAS G12C inhibitor except if ≥ 1 year has elapsed since last dose
3. Tumors harbouring other oncogenic drivers for which targeted therapy is available (note: patients with KRAS G12C mutation as a resistance mechanism on for example EGFR or ALK inhibitors are not eligible).
4. History of severe hypersensitivity reaction to JDQ443 or its excipients.
5. History of allogeneic bone marrow or solid organ transplant
6. Participant has had major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior to starting study treatment or has not recovered from side effects of such procedure.
7. Thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting the study treatment or participants who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs) radiotherapy ≤ 2 weeks prior to starting the study treatment or has not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting study treatment is allowed.
8. Clinically significant, uncontrolled cardiac disease and/or recent cardiac events (within 6 months), such as:

   * Unstable angina or myocardial infarction within 6 months prior to screening.
   * Symptomatic congestive heart failure (defined as New York Heart Association Grade II or greater).
   * Documented cardiomyopathy.
   * Clinically significant cardiac arrhythmias (e.g. sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker)
   * Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, unless controlled prior to first dose of study treatment.
   * History or current diagnosis of ECG abnormalities indicating significant risk of safety for study participation such as: concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker.
   * History of familial long QT syndrome or known family history of Torsades de Pointes.
   * Resting QT interval corrected with Fridericia's formula (QTcF) > 480 msec on screening ECG or congenital long QT syndrome.
   * Concomitant medication(s) with a "Known Risk of Torsades de Pointe" per www.qtdrugs.org that cannot be discontinued or replaced by safe alternative
9. A medical condition that results in increased photosensitivity (i.e. solar urticaria, lupus erythematosus, etc.).
10. History of interstitial lung disease or pneumonitis grade ≥ 2.
11. Current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (i.e. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes etc.).
12. Malignant disease, other than that is being treated in this study. Exceptions to this criterion include the following: malignancies that were treated curatively and have not recurred within two years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type.
13. Any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment cause unacceptable safety risks, contra-indicate participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, uncontrolled diabetes, hepatic disorders including cirrhosis).
14. Any other medical condition (such as active infection including known hepatitis or HIV, treated or untreated), which in the opinion of the Investigator represents an unacceptable risk for participation in the study.
15. Any medical condition or prior surgical resection that may affect the absorption of the investigational drug. Examples of medical conditions that may affect investigational drug absorption include (but are not limited to) inflammatory bowel disease (i.e. ulcerative colitis, Crohn's disease) and gastrointestinal disease such as ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, and malabsorption syndrome.
16. Participants who are taking a prohibited medication (strong CYP3A inducers) that cannot be discontinued at least seven days prior to the first dose of study treatment and for the duration of the study.
17. Use of any live vaccines against infectious diseases within four weeks of initiation of study treatment.
18. Participant is concurrently using other anti-cancer therapy.
19. Participation in any additional, parallel, investigational drug or device studies. Participation in non-interventional observational studies which will not influence the endpoints of the current studies is allowed (e.g. liquid biopsies, eNOSE, surveys).
20. Pregnant or breast-feeding women or women who plan to become pregnant or breast-feed during the study. Pregnant women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
21. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 7 days after the last dose of JDQ443.
22. Sexually active males unless they use a condom during intercourse while taking study treatment and for 7 days after the last dose of JDQ443. Male participants should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the study treatment via seminal fluid. In addition, male participants must not donate sperm and women participants must not donate oocytes for the time period specified above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
brain metastases overall response rate (ORR) | up to 24 months
  ORR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) based on central and local investigator's assessment according to RANO-BM criteria on brain MRI

SECONDARY OUTCOMES:
brain metastases disease controle rate (DCR) (key secondary) | up to 24 months
  DCR is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Non-CR/Non-PD according to RANO-BM on brain MRI
CNS progression free survival (PFS) (key secondary) | up to 24 months
  PFS is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS is based on local and central assessment according to RANO-BM on brain MRI
Extracranial ORR and DCR | up to 24 months
  ORR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) based on local investigator's assessment, DCR is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Non-CR/Non-PD according to RECIST 1.1, measured with CT
extracranial PFS | up to 24 months
  PFS is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS is based on local assessment according to RECIST 1.1 based on CT
overall PFS | up to 24 months
  median overall PFS based on RANO-BM for BM and RECIST 1.1 for extracranial lesions as defined above
overall survival | up to 33 months
  OS is defined as the time from date of start of treatment to date of death due to any cause
Change from baseline in EORTC QLQ-BN20 | up to 24 months
  the EORTC QLQ-BN20 is a questionnaire available that measures health-related quality of life of brain tumour patients
Change from baseline in EORTC QLQ-C30 | up to 24 months
  The EORTC QLQ-C30 is a questionnaire developed to assess the health-related quality of life of cancer participants
Safety according to CTCAE v5.0 | up to 24 months
  according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lizza Hendriks, MD, PhD, Principal Investigator — Maastricht University Medical Hospital

IPD SHARING:
Plan to Share IPD: No